CLINICAL TRIAL: NCT03272204
Title: Effects of Pubic Hair Grooming on Urinary and Vaginal Microbiome
Brief Title: Pubic Hair and the Urinary and Vaginal Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margaret Mueller (Other)
Responsible Party: Sponsor-Investigator, Margaret Mueller, Assistant Professor of Obstetrics and Gynecology, Urology, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00205206
Record Dates: First submitted 2017-08-18; First posted 2017-09-05 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: pubic hair; grooming; urinary tract symptoms; vaginitis
MeSH Terms: conditions — Grooming; Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Pubic Hair (Other): Participant with natural hair crosses over to removed pubic hair
  Interventions: Behavioral: No pubic hair
- Removed Pubic Hair (Other): Participant with no pubic hair crosses over to natural pubic hair
  Interventions: Behavioral: Pubic Hair

INTERVENTIONS:
Behavioral: No pubic hair — Natural pubic hair to fully removed pubic hair
  Arms: Natural Pubic Hair
Behavioral: Pubic Hair — Removed pubic hair to natural pubic hair
  Arms: Removed Pubic Hair

SUMMARY:
This research study seeks to find if there is a connection between the presence of pubic hair and the type of bacteria that live in the vagina and bladder.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are the most common bacterial infections. In 2007, in the United States alone, there were an estimated 10.5 million office visits for UTI symptoms (constituting 0.9% of all ambulatory visits) and 2-3 million emergency department visits. UTIs are significantly more common in women and are a leading cause of urogynecology referrals. In women, the vagina plays a key role in the pathogenesis of UTIs. The initial step in the pathogenesis of UTI is colonization of the vaginal opening and peri-urethra with uropathogens from the intestinal microbiota, followed by ascension of uropathogens via the urethra to the bladder and sometimes the kidneys to cause infection. Thus, understanding factors that affect the microbiota of the vagina is key to understanding the pathogenesis of UTI. Likewise, since Wolfe et al published the first evidence of a urinary microbiome in 2012, there has been growing interest in whether the content of this microbiome could correlate with symptoms of the lower urinary tract. The urinary microbiome has been shown to correlate with symptoms of urgency incontinence but to date, there is no data on whether the composition of the urinary microbiome is associated with any change in risk for UTIs. If the urinary microbiome could play a role in the acquisition of clinical infection, then the factors that affect the microbiome of the bladder would be important in preventing UTIs. One plausible and modifiable factor that may change the vaginal and urinary microbiome is the presence of pubic hair. Hair in other parts of the body (nose, ears, eyebrows) traps and stops the passage of pathogens into our mucous membranes. Additionally, the sebum produced by hair follicles is bacteriostatic. However, some form of pubic hair grooming is performed by the majority of pre-menopausal women (83%) and 62% of women between age 18-40 report having removed ALL of their pubic hair at one point in life. This is predominantly done by using non-electric razors (61%) but other women use lasers, waxing and depilatory creams. Fifty-nine percent of women who perform pubic hair removal report their primary reason is to improve hygiene. However, there is no data that this practice changes hygiene, with the exception of preventing pubic hair lice. On the contrary, pubic hair removal has been associated with skin injury leading to inoculation of bacteria and viruses. In a recent cross-sectional study of pubic hair and sexually transmitted infections, researchers found that frequent pubic hair grooming was correlated with a higher risk for sexually transmitted infections (STIs). This preliminary work raises the question of whether the presence of pubic hair affects the vaginal or urinary microbiome, thereby changing a woman's risk of infection in either organ. Furthermore, specific pelvic floor disorders (PFDs) including painful bladder syndrome and urgency urinary incontinence have been associated with specific microbiome profiles. Therefore, by falsely attempting to maintain pelvic health through grooming practices, women might inadvertently be exposing themselves to PFDs mediated by changes in their urinary or vaginal microbiomes. The aim of this study is to address this question through a pilot study of urinary and vaginal microbiomes in women with and without pubic hair AND in the same woman with and without pubic hair.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women between the ages of 18-50
* English-speaking
* Women with either natural growth/distribution of pubic hair or complete removal of pubic hair through a reversible process.
* Women who do not feel they have urinary or vaginal health problems and are not seeking care for these issues
* Women must be willing and able to complete study documentation and study procedures.

Exclusion Criteria: Women will be excluded for any of the following:

* Hair has been removed through an irreversible process like laser or electrolysis
* Patient feels they have bothersome urinary or pelvic floor conditions for which they are seeking care (for example: vaginal prolapse, frequent urinary incontinence, chronic pelvic pain, bladder pain)
* Patient plans on having any type of surgery in the next 2 months (due to likely antibiotic use)
* Patient has a history of a transplant and is on immunosuppression
* Patient has cancer for which she is currently getting chemotherapy or radiation
* Currently taking or has taken antibiotics in the last 7 days for any reason
* Patient has symptoms of a urinary tract or vaginal infection or is found on exam or culture to have a urinary tract infection or vaginal infection
* Patient is pregnant or breastfeeding
* Patient has douched in the last 48 hours
* Patient has had intercourse in the last 48 hours
* Patient is currently menstruating

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Comparison of Urinary and Vaginal Microbiomes | up to 3 months
  Describe and compare the urinary and vaginal microbiome in the same woman with natural pubic hair and with fully removed pubic hair

SECONDARY OUTCOMES:
Questionnaire Comparison | up to 3 months
  To compare questionnaire results for standardized patient surveys in the same woman with and without pubic hair
Self-Reported Infections | up to 3 months
  Comparing self-reported vaginal infections and urinary tract infections between women who have natural pubic hair and women who fully remove their pubic hair
Subtracting Microbiome Results | up to 3 months
  To suggest whether the transurethral urinary microbiome can be determined by subtracting the vaginal microbiome from the voided urinary microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Margaret G Mueller, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Geynisman-Tan J, Kenton K, Tavathia M, Yee A, Gilbert JA, Collins S, Lewicky-Gaupp C, Mueller M. Bare Versus Hair: Do Pubic Hair Grooming Preferences Dictate the Urogenital Microbiome? Female Pelvic Med Reconstr Surg. 2021 Sep 1;27(9):532-537. doi: 10.1097/SPV.0000000000000968. PMID 33181518